CLINICAL TRIAL: NCT02706392
Title: Phase I Study of Adoptive Immunotherapy for Advanced ROR1+ Malignancies With Defined Subsets of Autologous T Cells Engineered to Express a ROR1-Specific Chimeric Antigen Receptor
Brief Title: Genetically Modified T-Cell Therapy in Treating Patients With Advanced ROR1+ Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to slow accruals.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Maloney, Professor, Clinical Research Division, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9330; NCI-2015-01753 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9330 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9215045 (Other: Fred Hutch/University of Washington Cancer Consortium); 2R01CA114536 (NIH)
Record Dates: First submitted 2016-03-01; First posted 2016-03-11 (Estimated); Results first posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Triple-Negative Breast Carcinoma; Recurrent Acute Lymphoblastic Leukemia; Recurrent Mantle Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage III Lung Non-Small Cell Cancer AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7; Stage IV Lung Non-Small Cell Cancer AJCC v7; Unresectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Hematologic Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ROR1 CAR-specific autologous T-lymphocytes) (Experimental): Patients receive chemotherapy comprising fludarabine phosphate and cyclophosphamide as determined by the referring physician in consultation with the protocol PI. Beginning within 36-96 hours after completion of lymphodepleting chemotherapy, patients receive ROR1 CAR-specific autologous T-lymphocytes IV over 20-30 minutes. Patients may receive a second infusion of ROR1 CAR-specific autologous T-lymphocytes with or without additional cytoreductive therapy at the same (for those that received the highest cell dose) or up to the next highest dose level and there is persistent disease, there were no toxicities attributed to the first infusion, and the patient is at least 21 days from the first T cell infusion.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: ROR1 CAR-specific Autologous T-Lymphocytes

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: ROR1 CAR-specific Autologous T-Lymphocytes — Given IV
  Other Names: Autologous ROR1-CAR-T Cells; Chimeric Anti-ROR1 T-cell Receptor-expressing Autologous T-lymphocytes; ROR1-CAR-T

SUMMARY:
This phase I trial studies the side effects and best dose of genetically modified T-cell therapy in treating patients with receptor tyrosine kinase-like orphan receptor 1 positive (ROR1+) chronic lymphocytic leukemia (CLL), mantle cell lymphoma (MCL), acute lymphoblastic leukemia (ALL), stage IV non-small cell lung cancer (NSCLC), or triple negative breast cancer (TNBC) that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Genetically modified therapies, such as ROR1 specific chimeric antigen receptor (CAR) T-cells, are taken from a patient's blood, modified in the laboratory so they specifically may kill cancer cells with a protein called ROR1 on their surfaces, and safely given back to the patient after conventional therapy. The "genetically modified" T-cells have genes added in the laboratory to make them recognize ROR1.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of adoptive T cell therapy using ex vivo expanded autologous cluster of differentiation (CD)8+ and CD4+ ROR1 CAR-T cells for patients with advanced ROR1+ hematologic (Cohort A) and epithelial (Cohort B) malignancies.

SECONDARY OBJECTIVES:

I. To determine duration of in vivo persistence of adoptively transferred T cells, and the phenotype of persisting T cells.

II. To determine trafficking of adoptively transferred T cells traffic to the bone marrow or other tumor site and function in vivo.

III. To determine preliminary antitumor activity of the adoptive transfer of ROR1 CAR-T cells in patients with measurable tumor burden prior to T cell transfer.

OUTLINE: This is a dose escalation study of ROR1 CAR-specific autologous T-lymphocytes.

Patients receive chemotherapy comprising fludarabine phosphate and cyclophosphamide as determined by the referring physician in consultation with the protocol principal investigator (PI). Beginning within 36-96 hours after completion of lymphodepleting chemotherapy, patients receive ROR1 CAR-specific autologous T-lymphocytes intravenously (IV) over 20-30 minutes. Patients may receive a second infusion of ROR1 CAR-specific autologous T-lymphocytes with or without additional cytoreductive therapy at the same (for those that received the highest cell dose) or up to the next highest dose level and there is persistent disease, there were no toxicities attributed to the first infusion, and the patient is at least 21 days from the first T cell infusion.

After completion of study treatment, patients are followed up for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR PATIENTS WITH CLL, MCL OR ALL (COHORT A)

* CLL who are beyond first remission and who have failed combination chemoimmunotherapy with regimens containing a purine analogue and anti-CD20 antibody, or who have failed tyrosine kinase or phosphatidylinositol 3 (PI3) kinase inhibitors, or who were not eligible for or declined such therapy; patients with fludarabine refractory disease are eligible
* Mantle cell lymphoma patients who are beyond first remission and previously treated with chemoimmunotherapy; patients who have relapsed following autologous hematopoietic cell transplant (HCT) are eligible
* ALL patients who have relapsed or have residual disease following treatment with curative intent; ALL patients must have ROR1 expressed on > 90% of the leukemia blasts to be eligible
* Confirmation of diagnosis by internal pathology review of initial or subsequent biopsy or other pathologic material at the Fred Hutchinson Cancer Research Center (FHCRC)/Seattle Cancer Care Alliance (SCCA)
* Evidence of ROR1 expression by immunohistochemistry or flow cytometry on any prior or current tumor specimen
* Karnofsky performance status >= 70%
* Negative pregnancy test for women of childbearing potential; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Fertile male and female patients must be willing to use a contraceptive method before, during, and for at least two months after the T cell infusion
* Ability to understand and provide informed consent

INCLUSION CRITERIA FOR PATIENTS WITH NSCLC OR TNBC (COHORT B):

* Patients with non-small cell lung cancer that is metastatic or inoperable and who have been treated with at least one line of prior therapy or declined conventional therapy
* Patients with known epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) mutations must have been treated on at least one line of molecularly targeted therapy (e.g., erlotinib, crizotinib)
* Patients must have measurable disease by at least one of the criteria below:

  * Extra skeletal disease that can be accurately measured in at least one dimension as >= 10 mm with conventional computed tomography (CT) techniques as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
  * Skeletal or bone-only disease measurable by fludeoxyglucose F 18 (FDG) positron emission tomography (PET) imaging
* ROR1 expression in > 20% of the primary tumor or metastasis by immunohistochemistry (IHC)
* Karnofsky performance status of >= 70%
* Patients must be off chemotherapy for a minimum of 3 weeks prior to start of treatment; targeted therapies must be stopped at least 3 days prior to start of lymphodepletion
* Negative pregnancy test for women of childbearing potential; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Fertile male and female patients must be willing to use a contraceptive method before, during and for at least two months after the T cell infusion
* Ability to understand and provide informed consent

INCLUSION CRITERIA FOR TNBC:

* Histologically confirmed diagnosis of metastatic TNBC; i.e. breast cancer that is estrogen receptor (ER) negative (=< 10%), progesterone receptor (PR) negative (=< 10%), and human epidermal growth factor receptor 2 (HER2) negative (0 or 1+ by immunohistochemistry or negative for gene amplification by fluorescence in situ hybridization [FISH])
* Patients must have measurable disease by at least one of the criteria below:

  * Extra skeletal disease that can be accurately measured in at least one dimension as >= 10 mm with conventional CT techniques as defined by RECIST 1.1
  * Skeletal or bone-only disease measurable by FDG PET imaging
* Patients must have received standard adjuvant, neoadjuvant, and/or metastatic chemotherapy per National Comprehensive Cancer Network (NCCN) or institutional practice; no maximum on number of prior systemic treatment regimens
* Patients may receive agents to protect against skeletal related complications such as zoledronic acid or denosumab
* ROR1 expression in > 20% of the primary tumor or metastasis by IHC
* Karnofsky performance status of >= 70%
* Patients must be off chemotherapy for a minimum of 3 weeks prior to planned leukapheresis
* Negative pregnancy test for women of childbearing potential; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Fertile male and female patients must be willing to use a contraceptive method before, during and for at least two months after the T cell infusion
* Ability to understand and provide informed consent

Exclusion Criteria:

EXCLUSION CRITERIA FOR PATIENTS WITH CLL, MCL, OR ALL (COHORT A)

* Treatment with other investigational agent(s) within 30 days of planned lymphodepletion
* Patients requiring ongoing daily corticosteroid therapy at a dose of > 15 mg of prednisone per day (or equivalent); pulsed corticosteroid use for disease control is acceptable
* Active autoimmune disease requiring immunosuppressive therapy
* Serum creatinine > 2.5 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) > 5 x upper limit of normal
* Bilirubin > 3.0 mg/dL
* Patients with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing; those with a forced expiratory volume in 1 second (FEV1) of =< 65% or diffusion capacity of the lung for carbon monoxide (DLCO) (corrected) < 40% will be excluded
* Significant cardiovascular abnormalities as defined by any one of the following: congestive heart failure, clinically significant hypotension, symptomatic coronary artery disease, or a documented ejection fraction of < 45%; any patient with an ejection fraction (EF) of 45-49% must receive clearance by a cardiologist to be eligible for the trial
* Patients who are human immunodeficiency virus (HIV) seropositive
* Uncontrolled active infection (bacterial, viral, fungal, mycobacterial) not responding to treatment with intravenous antibiotics, antiviral or antifungal agents, or long-term treatment with oral agents
* Women who are breast-feeding
* Patients who have contraindication to cyclophosphamide chemotherapy
* Known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Untreated central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to enrollment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases

EXCLUSION CRITERIA FOR PATIENTS WITH NSCLC OR TNBC (COHORT B):

* Absolute neutrophil count (ANC) < 1000/mm^3
* Hemoglobin (Hgb) < 9 mg/dl (transfusion permitted to achieve this)
* Platelet count < 75,000/mm^3
* Treatment with other investigational agent(s) within 30 days of planned lymphodepletion
* Patients requiring ongoing daily corticosteroid therapy at a dose of > 15 mg of prednisone per day (or equivalent); pulsed corticosteroid use for disease control is acceptable
* Active autoimmune disease requiring immunosuppressive therapy
* Serum creatinine > 2.5 mg/dL
* SGOT > 5 x upper limit of normal
* Bilirubin > 3.0 mg/dL
* Patients with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing; those with an FEV1 of =< 65% or DLCO (corrected) < 40% will be excluded
* Significant cardiovascular abnormalities as defined by any one of the following: congestive heart failure, clinically significant hypotension, symptomatic coronary artery disease, or a documented ejection fraction of < 45%; any patient with an EF of 45-49% must receive clearance by a cardiologist to be eligible for the trial
* Patients who are HIV seropositive
* Uncontrolled active infection (bacterial, viral, fungal, mycobacterial) not responding to treatment with intravenous antibiotics, antiviral or antifungal agents, or long-term treatment with oral agents
* Women who are breastfeeding
* Patients who have contraindication to cyclophosphamide chemotherapy
* Known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Untreated central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to enrollment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases

EXCLUSION CRITERIA FOR TNBC:

* ANC < 1000/mm^3
* Hgb < 9 mg/dl (transfusion permitted to achieve this)
* Platelet count < 75,000/mm^3
* Treatment with other investigational agent(s) within 30 days of planned lymphodepletion
* Patients requiring ongoing daily corticosteroid therapy at a dose of > 15 mg of prednisone per day (or equivalent); pulsed corticosteroid use for disease control is acceptable
* Active autoimmune disease requiring immunosuppressive therapy
* Serum creatinine > 2.5 mg/dL
* SGOT > 5 x upper limit of normal
* Bilirubin > 3.0 mg/dL
* Patients with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing; those with an FEV1 of =< 65% or DLCO (corrected) < 40% will be excluded
* Significant cardiovascular abnormalities as defined by any one of the following: congestive heart failure, clinically significant hypotension, symptomatic coronary artery disease or a documented ejection fraction of < 45%; any patient with an EF of 45-49% must receive clearance by a cardiologist to be eligible for the trial
* Patients who are HIV seropositive
* Uncontrolled active infection (bacterial, viral, fungal, mycobacterial) not responding to treatment with intravenous antibiotics, antiviral or antifungal agents, or long-term treatment with oral agents
* Breast-feeding women
* Patients who have contraindication to cyclophosphamide chemotherapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Untreated central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to enrollment and any neurologic symptoms have returned to baseline) and have no evidence of new or enlarging brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osorio-Rodriguez DA, Camacho BA, Ramirez-Segura C. Anti-ROR1 CAR-T cells: Architecture and performance. Front Med (Lausanne). 2023 Feb 17;10:1121020. doi: 10.3389/fmed.2023.1121020. eCollection 2023. PMID 36873868
- [Derived] Srivastava S, Furlan SN, Jaeger-Ruckstuhl CA, Sarvothama M, Berger C, Smythe KS, Garrison SM, Specht JM, Lee SM, Amezquita RA, Voillet V, Muhunthan V, Yechan-Gunja S, Pillai SPS, Rader C, Houghton AM, Pierce RH, Gottardo R, Maloney DG, Riddell SR. Immunogenic Chemotherapy Enhances Recruitment of CAR-T Cells to Lung Tumors and Improves Antitumor Efficacy when Combined with Checkpoint Blockade. Cancer Cell. 2021 Feb 8;39(2):193-208.e10. doi: 10.1016/j.ccell.2020.11.005. Epub 2020 Dec 24. PMID 33357452

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A Dose Level 1: Patients with ROR1+ CLL, MCL or ALL that are refractory to conventional therapy will be eligible for Cohort A. Dose level 1 will be up to 3.3x105 EGFRt+ cells/kg. This is the starting dose for the study.
- Cohort A Dose Level 2: Patients with ROR1+ CLL, MCL or ALL that are refractory to conventional therapy will be eligible for Cohort A. Dose level 2 will be up to 1x106 EGFRt+ cells/kg.
- Cohort B Dose Level 1: Patients with ROR1+ NSCLC or TNBC who have failed conventional chemotherapy or targeted therapy, or for whom these therapies are not effective will be eligible for Cohort B. Dose level 1 will be up to 3.3x105 EGFRt+ cells/kg. This is the starting dose for the study.
- Cohort B Dose Level 2: Patients with ROR1+ NSCLC or TNBC who have failed conventional chemotherapy or targeted therapy, or for whom these therapies are not effective will be eligible for Cohort B. Dose level 2 will be up to 1x106 EGFRt+ cells/kg.
- Cohort B Dose Level 3: Patients with ROR1+ NSCLC or TNBC who have failed conventional chemotherapy or targeted therapy, or for whom these therapies are not effective will be eligible for Cohort B. Dose level 3 will be up to 3.3x106 EGFRt+ cells/kg.
- Cohort B Dose Level 4: Patients with ROR1+ NSCLC or TNBC who have failed conventional chemotherapy or targeted therapy, or for whom these therapies are not effective will be eligible for Cohort B. Dose level 4 will be up to 1.0x107 EGFRt+ cells/kg
Period: Overall Study
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
Started | 2 | 1 | 2 | 3 | 11 | 2
Completed | 1 | 1 | 0 | 1 | 6 | 0
Not Completed | 1 | 0 | 2 | 2 | 5 | 2
Not completed — Death | 1 | 0 | 2 | 2 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4 | Total
Number analyzed (Participants) | 2 | 1 | 2 | 3 | 11 | 2 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 2 | 2 | 7 | 2 | 14
  >=65 years | 1 | 1 | 0 | 1 | 4 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2 | 8 | 1 | 13
  Male | 2 | 1 | 0 | 1 | 3 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 2 | 3 | 9 | 0 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 2 | 3 | 9 | 2 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 2 | 3 | 11 | 2 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced Adverse Events
Description: Will be graded according to Common Terminology Criteria for Adverse Events. Outcome will be reported as a count of participants that experienced adverse events in each arm.
Time Frame: Within 35 days of receptor tyrosine kinase-like orphan receptor 1 positive chimeric antigen receptor-T cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
Number analyzed (Participants) | 2 | 1 | 2 | 3 | 11 | 2
Participants | 2 | 1 | 2 | 3 | 11 | 2

2. Secondary Outcome: Number of Participants With Persistence of Adoptively Transferred Receptor Tyrosine Kinase-like Orphan Receptor 1 Positive Chimeric Antigen Receptor-T Cells
Description: Data should be collected for persistence of transferred T cells and descriptive statistics will be used to summarize the changes from baseline where possible. This outcome is reported as a count of participants who experienced persistence at Day 28.
Time Frame: Up to 28 days after the T cell infusion
Population: Number analyzed is the number of participants that were evaluated for persistence in each arm. 2 patients were excluded because they went off study before their 1 month post treatment evaluation and were not assessed for persistence. 1 of these patients was in cohort A DL2. The other was in Cohort B DL4.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
Number analyzed (Participants) | 2 | 0 | 2 | 3 | 11 | 1
Participants | 2 | 0 | 2 | 1 | 0 | 0

3. Secondary Outcome: Number of Participants Biopsied With Detectable CD3 T-cells
Description: Samples of bone marrow, blood and other tissues (e.g. cerebral spinal fluid, tumor, thoracentesis fluid) will be collected from patients as clinically indicated. CD3 T-cells and their frequency/persistence will be detected by flow cytometry, polymerase chain reaction, and immunohistochemistry as appropriate. This outcome is reported as a count of participants who had detectable CD3 T-cells in their biopsy sample. The patients in Cohort A had a biopsy of their bone marrow. For the patients in Cohort B, biopsy location was dependent on site of disease per patient.
Time Frame: Up to 48 days post infusion
Population: Participants were analyzed if there was a biopsy done within 48 days post infusion. Biopsies were performed on 10 participants total, 2 participants in Cohort A and 8 participants in Cohort B.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
Number analyzed (Participants) | 2 | 0 | 2 | 3 | 3 | 0
Participants | 2 | 0 | 2 | 1 | 0 | 0

4. Secondary Outcome: Objective Response Rate of Complete Remission and Partial Remission
Description: Outcome will be reported as a count of participants in each arm that experienced complete remission and/or partial remission. For Patients with Acute lymphoblast leukemia (ALL), remission status will be determined by restaging of bone marrow and other involved sites by morphology, flow cytometry and molecular studies, as appropriate. For Patients with NSCLC and TNBC, tumor response and progression will be evaluated in this study using the international criteria proposed by RECIST Criteria. Target lesion responses will be described as (1) Complete response (CR): disappearance of all target lesions; (2) Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and, (4) Stable Disease: neither sufficient shrinkage to qualify for PR nor sufficient growth to qualify for PD.
Time Frame: Up to 1 year
Population: In arm 1, one patient was not assessed for a response and therefore is not included in the "number of participants analyzed" count.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 11 | 2
Participants | 0 | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Progression Free Survival
Description: Outcome will be reported as a count of participants in each arm that survived up to 1 year post-infusion (per patient) and did not progress. For patients with Acute lymphoblast leukemia (ALL), remission status will be determined by restaging of bone marrow and other involved sites by morphology, flow cytometry and molecular studies, as appropriate. For Patients with NSCLC and TNBC, tumor response and progression will be evaluated in this study using the international criteria proposed by RECIST Criteria. Target lesion responses will be described as (1) Complete response (CR): disappearance of all target lesions; (2) Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and, (4) Stable Disease: neither sufficient shrinkage to qualify for PR nor sufficient growth to qualify for PD.
Time Frame: Up to 1 year
Population: Only participants that survived up to 1 year post-infusion (per patient) could be analyzed for this outcome. In arm 1, one patient survived up to 1 year but they were not assessed for a response, therefore are not included in the "number of participants analyzed" count.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 6 | 0
Participants | 0 | 0 | 0 | 0 | 1 | 0

6. Secondary Outcome: Overall Survival
Description: Data should be collected for efficacy of transferred T cells and descriptive statistics will be used to summarize the changes from baseline where possible. Outcome will be reported as a count of participants that survived up until the 1 year post-infusion (per patient) timepoint.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
Number analyzed (Participants) | 2 | 1 | 2 | 3 | 11 | 2
Participants | 1 | 1 | 0 | 1 | 6 | 0

ADVERSE EVENTS:
Time Frame: Up to one year following last infusion per patient
Description: The NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4 was used for grading and analysis of adverse events. All grade 3 or greater adverse events were collected from time of leukapheresis until commencement of new anti-tumor therapy or until one year post infusion, whichever came first.
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/1 | 2/2 | 2/3 | 5/11 | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/1 | 1/2 | 2/3 | 10/11 | 2/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 2/2 | 3/3 | 11/11 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Dose Level 1 (N=2) | Cohort A Dose Level 2 (N=1) | Cohort B Dose Level 1 (N=2) | Cohort B Dose Level 2 (N=3) | Cohort B Dose Level 3 (N=11) | Cohort B Dose Level 4 (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 9 (12) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Dose Level 1 (N=2) | Cohort A Dose Level 2 (N=1) | Cohort B Dose Level 1 (N=2) | Cohort B Dose Level 2 (N=3) | Cohort B Dose Level 3 (N=11) | Cohort B Dose Level 4 (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 5 (6) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (15) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 3 (6) | 11 (13) | 1 (4)
Neutrophil count decreased (Investigations) | 2 (3) | 1 (4) | 2 (2) | 3 (6) | 11 (11) | 1 (1)
Platelet count decreased (Investigations) | 2 (4) | 1 (1) | 0 (0) | 1 (2) | 4 (4) | 1 (1)
White blood cell decreased (Investigations) | 2 (4) | 1 (2) | 2 (2) | 3 (6) | 11 (12) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Hypertension (Vascular disorders) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT02706392/Prot_SAP_000.pdf